CLINICAL TRIAL: NCT00570557
Title: Development of a Web-Based Course to Maintain Skills in Nurses Trained to Screen for Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06354
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Deglutition Disorders; Dysphagia; Stroke
Keywords: Skill Maintenance; Skill Decay; Screening
MeSH Terms: conditions — Deglutition Disorders; Stroke

ARMS (2):
- Group A Nurses (No Intervention): Participants receive neither web-based refresher courses nor periodic feedback by SLP
- Group B Nurses (Experimental): Participants receive web-based skill refresher courses but no periodic feedback by SLP
  Interventions: Other: TOR-BSST© Refresher Training

INTERVENTIONS:
Other: TOR-BSST© Refresher Training — Web-based refresher training in dysphagia screening
  Arms: Group B Nurses

SUMMARY:
This research aims to facilitate the successful implementation of the new Heart and Stroke Foundation of Ontario dysphagia screening model for acute stroke patients. The objectives will be 1) to determine the natural history of dysphagia screening skill decay, and 2) to assess the benefit of independent web-based practice and periodic feedback on screening skill maintenance. We will enrol a convenience sample of nurses who currently work with stroke patients but who have had no prior formal training with dysphagia screening.

The study will consist of 2 phases: A) an initial pilot phase followed by B) a prospective randomized controlled study. During Phase A, three new web-based, self-instructed skill refresher courses will be developed to help nurses maintain the skills they will learn in an 8-hour workshop on dysphagia screening. During Phase B, nurses will receive the 8-hour workshop and one-on-one evaluation by a speech-language pathologist (SLP). Following training, competent screeners will be randomized into one of two groups: Group A - Control group with no refresher course or periodic feedback from SLP; Group B - Web-based skill refresher courses only. Nurses will be evaluated at several timepoints throughout Phase B to assess theoretical dysphagia screening knowledge and skills.

ELIGIBILITY:
Inclusion Criteria:

* Nurses who care for acute stroke patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2007-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Skill decay over time among nurses trained to use the TOR-BSST© to screen for dysphagia in stroke patients | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary Martino, MA, MSc, PhD, Principal Investigator — University of Toronto, Dept. of Speech Language Pathology
Locations (5):
- Our Lady of Lourdes Hospital, Binghamton, New York, United States
- Canada (4):
  - Foothills Hospital, Calgary, Alberta
  - Alberta Health Services - Capital Health (University of Alberta Hospital, Royal Alexandra Hospital), Edmonton, Alberta
  - Georgian Bay General Hospital, Penetanguishene/Midland, Ontario
  - University Health Network - Toronto Western Hospital, Toronto, Ontario

REFERENCES:
- [Background] Martino R, Foley N, Bhogal S, Diamant N, Speechley M, Teasell R. Dysphagia after stroke: incidence, diagnosis, and pulmonary complications. Stroke. 2005 Dec;36(12):2756-63. doi: 10.1161/01.STR.0000190056.76543.eb. Epub 2005 Nov 3. PMID 16269630
- [Background] Martino R, Pron G, Diamant N. Screening for oropharyngeal dysphagia in stroke: insufficient evidence for guidelines. Dysphagia. 2000 Winter;15(1):19-30. doi: 10.1007/s004559910006. PMID 10594255
- [Background] Martino R, Silver F, Teasell R, Bayley M, Nicholson G, Streiner DL, Diamant NE. The Toronto Bedside Swallowing Screening Test (TOR-BSST): development and validation of a dysphagia screening tool for patients with stroke. Stroke. 2009 Feb;40(2):555-61. doi: 10.1161/STROKEAHA.107.510370. Epub 2008 Dec 12. PMID 19074483
- See also: Swallowing Lab Website — http://swallowinglab.uhnres.utoronto.ca